CLINICAL TRIAL: NCT05171985
Title: Dexmedetomidine Sedation Reduces Atrial Fibrillation in Mechanically Ventilated Patients With COVID-19 Pneumonia: a Randomized Controlled Trial
Brief Title: Dexmedetomidine Reduces Atrial Fibrillation in Mechanically Ventilated Patients With COVID-19 Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amr Arafa Elbadry, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dexmedetomidine sedation
Record Dates: First submitted 2021-12-20; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: COVID-19 Pneumonia; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine sedation group (Experimental): 72 cases sedated on Propofol infusion 50-200 mg/h + Fentanyl infusion 25-250 mcg/h guided by hemodynamics in addition to Dexmedetomidine infusion 0.2 - 1 mcg/kg/h, and also guided by hemodynamics.
  Interventions: Procedure: Dexmedetomidine sedation
- control group (Other): 72 cases sedated on Propofol infusion 50-200 mg/h + Fentanyl infusion 25-250 mcg/h guided by hemodynamics
  Interventions: Procedure: Dexmedetomidine sedation

INTERVENTIONS:
Procedure: Dexmedetomidine sedation — 72 cases sedated on Propofol infusion 50-200 mg/h + Fentanyl infusion 25-250 mcg/h guided by hemodynamics in addition to Dexmedetomidine infusion 0.2 - 1 mcg/kg/h, and also guided by hemodynamics.

SUMMARY:
Coronavirus disease 2019 (COVID-19) is a novel, has rapid spread worldwide. Currently, almost 11 million cases have been diagnosed and more than 500,000 infected people have died rather than undiagnosed patients .

Although COVID-19 is mostly characterized by the respiratory tract affection, cardiovascular complications frequently accompany COVID-19 infections increasing morbidity and mortality in such patients .

Arrhythmias are frequently reported in COVID-19 patients, with atrial fibrillation (AF) being the most common form . Although electrical, calcium handling, and structural remodeling plays a key role in AF pathophysiology , the clinical presentation of AF is diverse and the precise mechanisms of AF remain unclear in this large proportion of patients .

In patients with severe pneumonia, acute respiratory distress syndrome (ARDS) and sepsis, the incidence of AF during hospitalization is usually high . For instance, about 23-33% of critically ill patients with sepsis or ARDS have AF recurrences and 10% develop de novo AF.

Dexmedetomidine preserves the natural sleep pattern and induces cooperative sedation in which patients are easily arousable, leading to to less impairment in cognitive function. In addition, it has an opioid sparing effect, and it is associated with a significant decrease in the duration of delirium, ventilatory care along with ICU stay, and therefore it is associated with a significant improvement in outcomes. These mentioned advantages make dexmedetomidine a fundamental sedative in ICU practice .

The use of dexmedetomidine to prevent atrial fibrillation is unclear . However, two retrospective studies also showed that dexmedetomidine sedation might

DETAILED DESCRIPTION:
All cases will be commenced on invasive mechanical ventilation pressure-controlled ventilation on peak end expiratory pressure (PEEP) ≥ 10 cmH2O, inspiratory pressure (Pi) adjusted to keep plateau pressure less than 30 cmH2O, respiratory rate set between 20 and 35 keeping PH more than 7.15 The included cases will be randomized using the closed envelope method into two groups; Group I will include 72 cases sedated on Propofol infusion 50-200 mg/h + Fentanyl infusion 25-250 mcg/h guided by hemodynamics, whereas Group II will include the remaining 72 cases who will be sedated using the same regimen of group I in addition to Dexmedetomidine infusion 0.2 - 1 mcg/kg/h, and also guided by hemodynamics.

The incidence of AF will be monitored and recorded. AF will be defined as a supraventricular arrhythmia characterized by disorganized atrial depolarization without effective atrial contractions. If AF terminates spontaneously, it is defined as paroxysmal. When AF is sustained beyond seven days or is terminated with electrical or pharmacological cardioversion it is defined as persistent. If a conversion in sinus rhythm cannot be achieved, AF is defined as permanent (24). Also, Troponin level every 8 hours and ECG 3 times all over the day of AF episode.

Management of the attacks of rapid AF will be as follow; in hemodynamically unstable patients, synchronized external direct-current cardioversion will be performed with the pads placed anteriorly and posteriorly (over the sternum and between the scapulae) at 100 joules (J). If no response occurs, the current will be applied again at 200 J; if there is still no response, the current will be increased to 300 J, and then to a maximum of 360 J.

If patients cannot be moved, the pads will be applied over the right sternal border and left lateral chest wall .

In hemodynamically stable patients, amiodarone will be given; with a loading dose of 300 mg iv infusion over 30 min, then a maintenance dose 900 mg iv infusion over 24 hours with monitoring of blood pressure. Metoprolol 25-50 mg tablets bd will be added to the medication list provided hemodynamic stability .

The number of AF attacks in each group will be our primary outcome. Secondary outcomes will include number of cases requiring cardioversion and incidence of mortality.

Measurements:

1. Number of attacks of AF in each group.
2. Number of DC shocks.
3. Total dose of amiodarone.
4. Total dose of metoprolol.
5. Incidence of mortality in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥18 years
* confirmed to have COVID-19 pneumonia by nasopharyngeal swab PCR together with chest radiology
* requiring invasive mechanical ventilation.

Exclusion Criteria:

* heart rate <50 beats per minute,
* atrioventricular conduction block of grade II or III,
* mean arterial pressure (MAP) <55 mmHg (despite appropriate intravenous volume replacement and vasopressor treatment),
* acute severe neurological disorder,
* propofol or dexmedetomidine allergy or other contraindications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The number of atrial fibrillation (AF) attacks | one month
  The number of atrial fibrillation (AF) attacks in each group will be our primary outcome

SECONDARY OUTCOMES:
1) Number of DC shocks | one month
  Number of DC shocks
2) Total dose of amiodarone | one month
  Total dose of amiodarone
3) Total dose of metoprolol | one month
  Total dose of metoprolol

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ELgharbiaa, Egypt